CLINICAL TRIAL: NCT03781076
Title: Sleep After Adolescent Mild Traumatic Brain Injury (mTBI, Aka Concussion): Nature, Contributors, and a Pilot Clinical Trial
Brief Title: Sleep After Adolescent Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cincinnati Children's Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB number 2018-5952
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Brain Concussion
Keywords: Adolescence, Sleep
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Note that the intervention portion of the study involves only a subset of participants. The larger bulk (planned n=108) will undergo only initial observation of sleep and concussion symptoms. The investigators plan to have 24 (those still symptomatic at 4 weeks post-concussion who do not get recommended sleep) undergo a pilot trial of a sleep intervention.
Who Masked: Outcomes Assessor
Masking Description: The intervention explicitly involves behavior change, so the participant cannot be blinded. The outcomes assessment involves objective monitors, and therefore can be considered blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Intervention (Experimental): 1-hour brief behavioral intervention to improve sleep consolidation and nocturnal sleep duration.
  Interventions: Behavioral: Sleep Intervention
- Control (No Intervention): In this "care as usual" arm, no specific behavioral sleep intervention is provided.

INTERVENTIONS:
Behavioral: Sleep Intervention — The study therapist will outline the biopsychosocial model of mTBI recovery, highlighting the shift from biological injury to behavior (especially sleep behavior) as key driver of symptoms. The intervention will then apply well-established strategies from the pediatric psychology and insomnia literatures, encouraging conjoint problem-solving by parent and youth with the shared goal of maximizing nocturnal sleep. These include: pre-planning, problem-solving, development of a positive routine, commitment to sleep-promoting behaviors, self-monitoring, and positive reinforcement. The therapist will also teach a brief, self-guided pre-sleep relaxation exercise that has been used in insomnia treatment to maximize the benefit of additional sleep opportunity.
  Arms: Sleep Intervention

SUMMARY:
The purpose of this research study is to learn more about how sleep changes as teens recover from concussions. We also want to learn if we can improve sleep in teens who have concussions.

DETAILED DESCRIPTION:
Mild traumatic brain injuries (mTBI), also called concussions, affect millions of individuals and cost over $17 billion in the US annually. Despite the term "mild," mTBI symptoms in children and adolescents (e.g., poor concentration, headache, emotional lability, slow thinking) seriously disrupt all aspects of a patient's functioning and impair quality of life. Although many youth recover quickly from mTBI, 30-60% remain symptomatic a month later. A biopsychosocial model was developed to account for protracted recoveries. In this model, acute symptoms result from a rapid cascade of injury-related neurometabolic and micro-structural aberrations. Since the vast majority of these abate within 1-3 weeks post-injury, persistent symptoms become increasingly difficult to explain physiologically, and psychosocial circumstances and patient behaviors become increasingly prominent contributors to impairment. There is reason to believe that, after mTBI, sleep is an underappreciated, modifiable behavior that drives impairment for youth with protracted recoveries. Care recommendations often mention sleep, but the field lacks empirically-supported guidelines and interventions for sleep after pediatric mTBI. Studies of mTBI in youth have used crude, unvalidated sleep measures. Also, there is no systematic research on non-injury contributors to poor sleep after mTBI, nor the nature and sources of advice that families receive. Lacking such data, one cannot develop empirically-based sleep recommendations. Finally, while there is reason to believe that a brief sleep intervention can alleviate mTBI symptoms in many youth who are recovering slowly, this needs to be tested in a well-powered clinical trial. The investigators are positioning to undertake such a trial, but must first document feasibility and acceptability of a sleep intervention after mTBI. To address these research gaps, the investigators are conducting a novel observational study and pilot clinical trial with these Aims:

Aim 1: Establish more detailed and definitive links between protracted mTBI recovery and sleep in 12-18-year-olds. The investigators are undertaking a prospective, observational study, objectively tracking sleep and assessing recovery 3-4 weeks post-mTBI. The study team will also explore potential contributors to inadequate sleep, including sleep-related behaviors and detail the nature and sources of information on sleep post mTBI.

Aim 2: Pilot-test a brief sleep intervention in the subset of youth who are slow to recover from mTBI and show short sleep. The study team will document feasibility and acceptability, and test its success in extending sleep duration.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old
* Had a mild TBI or concussion (blow to the head associated with loss of consciousness<30 min, amnesia, or alteration in mental status) <3 weeks prior to study participation.

Exclusion Criteria:

* lowest Glasgow coma scale (GCS) <13 or imaging evidence of intracranial abnormality (i.e., too severe)
* previous more severe TBI or mTBI within the prior 3 months (potential overlapping recoveries)
* extracranial injury with an Abbreviated Injury Severity Scale >4 for that region (non-mTBI injuries)
* non-fluent in English
* previously-diagnosed intellectual disability, autism, bipolar disorder, or psychosis (could impact measure validity)
* use of medication known to substantially affect sleep (e.g., stimulant).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep | 1-2 weeks
  Nocturnal sleep duration, quality, and regularity, as measured by wrist-mounted accelerometry (actigraphy). Although in theory there are upper limits on healthy sleep, in practice during adolescence better health is associated with longer nocturnal sleep, better sleep quality, and greater night-to-night consistency in sleep patterns.
Concussion Symptoms | 1-2 weeks
  A primary outcome for the observational phase of the study, and a secondary outcome for the intervention phase, will be the Post-Concussion Symptom Scale (PCSS). On the PCSS, 21 common symptoms after concussion are rated on a 0-6 scale; for this study the focus will be on the summed total across items. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Dean W Beebe, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
A deidentified data set may be available to qualified researchers who share specific research idea with the central contact person (Dr. Beebe, PI).